CLINICAL TRIAL: NCT06408779
Title: Study on Surgical Treatment Strategies for Moderate Ischemic Mitral Regurgitation
Status: Completed | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: m_IMR_2024
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Mitral Valve Insufficiency; Mitral Valve Annuloplasty; Coronary Artery Bypass
MeSH Terms: conditions — Mitral Valve Insufficiency | interventions — Mitral Valve Annuloplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- coronary artery bypass grafting
  Interventions: Procedure: mitral valve repair
- coronary artery bypass grafting concomitant mitral valve repair
  Interventions: Procedure: mitral valve repair

INTERVENTIONS:
Procedure: mitral valve repair — coronary artery bypass grafting concomitant mitral valve repair

SUMMARY:
This study aimed to compare the efficacy of isolated coronary artery bypass grafting and coronary artery bypass grafting + mitral valve repair in moderate ischemic mitral regurgitation patients through a cohort and explore the potential risk factors of the clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Adult coronary artery disease patients complicated with moderate ischemic mitral regurgitation.
2. undergoing coronary artery bypass grafting with or without mitral valve repair.

Exclusion Criteria:

1. patients under the age of 18 years,
2. patients complicated with more than moderate ischemic mitral regurgitation or undergoing mitral valve replacement,
3. patients complicated with primary mitral valve disease other than ischemic mitral regurgitation, such as rheumatic mitral regurgitation or mitral valve leaflet prolapse,
4. patients undergoing concomitant aortic valve procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult coronary artery disease patients complicated with moderate ischemic mitral regurgitation undergoing coronary artery bypass grafting with or without mitral valve repair from August 2009 to August 2023 were enrolled
Sampling Method: Non-Probability Sample
Enrollment: 464 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
major adverse cardiovascular and cerebrovascular events | 2years
  the composite of all-cause death, rehospitalization for heart failure, non-fatal myocardial infarction, non-fatal stroke or repeat mitral valve surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China